CLINICAL TRIAL: NCT04561167
Title: Clinical Performance of the Indirect Resin Composite Restorations in Endodontically Treated Teeth With Different Cavity Preparation Designs: (A Randomized Clinical Trial)
Brief Title: Clinical Performance of the Indirect Resin Composite Restorations in Endodontically Treated Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hoda omar tawfeek hussien fouda, The principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Egameel43
Record Dates: First submitted 2020-09-13; First posted 2020-09-23 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cuspal reduction in MOD Cavity in endodontically treated teeth (Experimental): Cavity design is of prime importance for the restoration of endodontically treated teeth. The cavity design plays an important role in the protection of the remaining tooth structure as well as the restoration. Cuspal reducuction and further coverage by the CAD/CAM generated indirect resin composite restoration has been proved in literature by the retrospective study done by (Chrepa V et al 2014) which studied 189 posterior endodontically treated teeth receiving indirect composite onlays with a median follow up time of 37 months and suggested this type of restoration as a viable option with 100% tooth survival and 96.8% restoration survival.
  Interventions: Other: Cuspal reduction in MOD cavity in endodontically treated teeth
- No cuspal reduction in endodontically treated teeth (Active Comparator): In the present study, choosing the comparator to be the cavity design without cuspal reduction and further coverage (inlay) is done as an attempt to reduce the application of inlays in endodontically treated teeth. In accordance to the in-vitro study done by (M. D. Al Amri et al 2016) which tested the fracture resistance of endodontically treated mandibular first molars with conservative access cavity and different restorative techniques, catastrophic failures were highest in the composite group (100%), followed by the inlay and the amalgam groups (91.67%) and this was referred to the adhesive bonding mechanism of the composite restoration and the wedging effect of the inlay and the amalgam restorations (Rivera EM andWalton RE 2015)
  Interventions: Other: No cuspal reduction in MOD cavity in endodontically treated teeth

INTERVENTIONS:
Other: Cuspal reduction in MOD cavity in endodontically treated teeth — Not only the quality of endodontic treatment that affects the prognosis of the endodontically treated tooth, but the subsequent restorative treatment as well. Coverage, Endocrowns, Onlays, Inlays Restorations on Fracture Resistance of Endodontically Treated Molars, it was found that the worst results came to the inlay restorations and this was attributed to geometric form of preparation that exert a wedging force acting to split the tooth when under occlual stress however, onlay and full coverage direct the force along the long axis by overlaying the cusp tips and a portion of buccal and lingual surface thus opposing the wedging action created by internal design of restoration (Magne P and Belser C. et al 2003) That's why, choosing such a design as a comparator to the design of the cuspal reduction and further coverage (onlay) is crucial to show the importance of cuspal coverage for the indirect resin composite restoration in the endodontically treated teeth.
  Arms: Cuspal reduction in MOD Cavity in endodontically treated teeth
Other: No cuspal reduction in MOD cavity in endodontically treated teeth — In an invitro study done by (Ahmed Hamdy 2015) investigating the effect of Full The amount of lost internal tooth structure as well as the coronal hard tissue in an endodontically treated tooth is considered the main factors that make the tooth susceptible to biomechanical failure when compared to a vital tooth. (Guo J et al 2016) .
  Arms: No cuspal reduction in endodontically treated teeth

SUMMARY:
Does the cuspal reduction during cavity preparation for indirect resin composite restorations in endodontically treated teeth increase the clinical performance when compared to cavities prepared without cuspal reduction?

DETAILED DESCRIPTION:
Selection and examination of the all patients will be done according to inclusion and exclusion criteria( by Hoda omar fouda in the Faculty of Dentistry Cairo University, Egypt ) from the outpatient clinic of the conservative department of the faculty of oral and dental medicine , cairo university .Patients should have an endodontically treated molar with remaining three walls fulfilling the inclusion criteria of the selected teeth or patients who need root canal treatment to be done prior to restoration to be enrolled in the study. Root canal treatment for all patients will be done by step back technique using rotary files .Sodium hypochlorite and EDTA solution will be used as root canal irrigant solution. Root canals will be obturated with gutta percha cones using AH Plus (Dentsply, Konstanz Germany). Eugenol based sealers will avoided to avoid the contamination of the remaining walls with eugenol that can interfere with the polymerization of the adhesive.

Eugenol free temporary filling material (Coltosol F by Coltene, Switzerland) will be used to seal the cavity till the restorative visit A digital periapical radiograph will be done to check the quality of the root canal treatment. The selected tooth should be free from any periapical radiolucency, missed canals or poor obturation. The periodontal condition of the tooth will be also checked radiographically. The tooth should be free from any clinical symptoms as pain on biting or swelling. A period not more than a month should pass from the root canal treatment to avoid any coronal leakage that might affect the prognosis of the root canal treatment during the time of the study. Any defects in the temporary filling material should be restored again to assure proper coronal seal till the beginning of the treatment. Before the removal of the temporary filling, assessment of centric and eccentric occlusal contacts will be performed with an articulating paper. The tooth should be then checked for the contact points in the centric relation and eccentric movements It is important to determine the contact points during the centric and eccentric movements to maintain the tooth restoration interface at a stress free areas as much as possible for more durable bonding. The quadrant with the cavity will be isolated using rubber dam system with two suctions tips one below the rubber dam sheet and the other one near to the tooth to keep the working area always clean and keep the patient comfortable during the procedures. Using straight and round blue coded diamond stones attached to high speed handpiece with copious air and water coolant, the temporary filling will be removed from the cavity. The cavity should then be checked for any remaining carious lesions to be removed. All the undermined enamel walls should be removed so that all the remaining cavity walls have well supported sound enamel margins. Any soft carious lesions will be by a sharp spoon excavator. Any gutta-percha remnants in the pulp chamber should be removed till the gutta percha becomes at the level of the orifice and all the walls and floor are completely clean. All the procedures will be performed with magnifying loupes 3.5 x (Univet, Italy). The angulation of the cavity walls will be adjusted to be 6 degrees diverge of the axial inclination using blue coded diamond tapered with round end bur diameter 16, length 10.

Standardization of the prepared cavity dimensions should be done as follows:

1. For the inlay group thickness of remaining walls (in order to maintain them) has to be 1.5 mm.
2. The occlusal inter-cuspal distance ranges from 4-5 mm

4- Width of occlusal isthmus had to be 2-3 mm. 5- Buccal and lingual walls of the proximal parts of the cavity will be prepared using the same diamond bur (MIDWEST Dentsply) used for the occlusal part of the cavity to provide the same angle of divergence (6 degrees) as that of the occlusal walls. 6- The proximal boxes corresponds to one-third the distance between the buccal and lingual surfaces of the teeth 7- The gingival floor of the proximal part of the cavity has to be continuous with the pulpal floor of the occlusal part having the same depth. 8- Interproximal overjet has to be ≤ 2 mm. 9- The internal line angles should be rounded, the cavo-surface angles should be 90° For the Intervention Group: no cuspal reduction will be done as these will be the cavities prepared to receive the inlay restorations For the Comparator Group: cuspal reduction to buccal and lingual cusps will be done as these will be the cavities prepared to receive the onlay restorations

Acid etching:

Selective etching technique using a 35% phosphoric acid gel (Scotchbond™ Universal Etchant 3M) on the marginal enamel for 15 seconds. The gel will then thoroughly rinsed for about 30 seconds using air water spray and then air dried for 5 seconds.

Application of adhesive:

After proper dryness and with the aid of a micro-brush (Microbrush International, USA), the Prime and Bond universal adhesive (Dentsply Sirona) will be applied over all the cavity surfaces according to the manufacturer's instructions and rubbed for 20 seconds then blown with a gentle air blow for 5 seconds to evaporate the solvent and then light cured for 10 seconds using LED curing light (Elipar S10, 3M ESPE) at a light intensity of 1200 mw/cm2.

Application of the base:

Bulk fill flowable composite SDR (Dentsply sirona) of universal shade will be directly applied to the floor of the cavity to fill the pulp chamber from bottom to top and light cured for 10 seconds according to the manufacturer's instructions with the same light curing device as the adhesive.

Milling of the designed restoration:

The operator will adhere strictly to the manufacturer's instructions in the imaging, computer design and machining of the restorations. A CEREC Primescan unit with Operating System 1.21 and the extended machining option for the milling process. BRILLIANT Crios Composite Blocks for CEREC® will be used to design and mill the inlays and onlays.

Cementation protocol:

The fitting surface of the restoration will be treated as follows to be ready for cementation:

* Sandblasting by AquaCare Air Abrasion Unit using aluminum oxide particles of 0.5 mm particle size.
* Ultrasonic cleaning using InvisiClean ultrasonic cleaner for one minute.
* Prime and bond universal adhesive layer will be applied, air thinned for 5 seconds and cured for 10 seconds The RelyX Unicem clicker 3M ESPE will be used for the restoration cementation and final finishing and polishing will be done if any occlusal adjustments are done to the restoration

ELIGIBILITY:
Inclusion Criteria:

* Only co-operative patients approving to participate in the trial.
* Good oral hygiene.
* Medically free adult patients.
* The age range of the patients is 13-18 years
* Patients havind Endodontically treated molars with remaining two walls.
* Teeth with no periapical lesion or radiolucency.
* Root canal treatment finished from maximum two weeks with no clinical symptoms.
* Prepared cavity with no undermined enamel walls.
* The thickness of the remaining walls not less than 2 mm.
* Functioning tooth with presence of an opposing.
* Healthy periodontium

Exclusion Criteria:

* Old age patients.
* Patients with disabilities.
* Patients having systemic diseases or severe medically compromised.
* Patients with of severe bruxism, clenching or temporomandibular joint disorders.
* Poor oral hygiene.
* Teeth with severe dilacerations.
* Teeth with periapical lesions.
* Teeth with visible cracks.
* Teeth with internal or external root resorption.
* Teeth with calcified root canals.
* Teeth with mobility.
* Teeth with undermined enamel walls.
* Non-functioning tooth with no opposing tooth.
* Heavy occlusion or signs of severe attrition.
* Severe periodontal affection.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Marginal adaptation | 12 months
  Visual inspection with explorer and mirror by measuring the distance penetrated by the explorer at the tooth restoration interface.
  The explorer will be drawn across the surface of the restoration toward the tooth

SECONDARY OUTCOMES:
Fracture of tooth and /or restoration | 12 months
  Visual inspection with explorer and mirror, to find the amount of fracture either in tooth or restoration
Anatomic Form | 12 months
  Degree of Continuity between natural tooth structure and the restoration
  Tactile sensation checking the anatomic form to show if there is no discontinuity, slight discontinuity or discontinuity and failure
Surface texture | 12 months
  Area of continuous movement of an explorer across the surface of the restoration
  Surface texture is highly polished or gritty containing supramicron-sized particles or Surface pitting is coarse to inhibit the continuous movement of an explorer across the surface
post operative sensitivity | 12 months
  Pain due to dentin hypersensitivity (evaporative stimulus)
  Pain arising from dentin hypersensitivity around the restoration stimulated by air blast measured by YES or NO scale
Retention | 12 months
  Visual inspection by the explorer and mirror to find out if there is loss of the restoration or no loss of the restoration
Color Match | 12 months
  The degree of mismatch from the normal range of tooth shades and translucency
  Visual inspection to check the proximity of the shade from the natural tooth
Secondary Caries | 12 months
  Distance penetrated due to secondary caries by visual evidence of dark keep discoloration adjacent to the restoration but not directly associated with cavosurface margins
  Visual inspection of discoloration that occurs on the tooth after the filling has been used for a period of time

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Fouda, master, Principal Investigator — Cairo University
Locations (1):
- Hoda omar fouda, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Undecided: It is not yet known if there will be a plan to make IPD available.
Supporting Information: Study Protocol
Time Frame: expecting to have all the data during october 2022
Access Criteria: IPD through contacting the main author Hoda.fouda@bue.edu.eg
URL: http://erepository.cu.edu.eg/index.php/cutheses